CLINICAL TRIAL: NCT06845761
Title: Examining the Relationship Between Ongoing Alcohol Use, Suicidal Thoughts and Behaviors and Related Constructs, and Behavioral Economic Decision-Making
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mark J Rzeszutek, PhD (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Mark J Rzeszutek, PhD, Post Doctoral Scholar, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 97418; K99AA031309-01A1 (NIH)
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Use; Suicidal Ideation/Behavior
Keywords: Alcohol; Cognitive Behavioral Therapy; Suicide; Remote; Self-Guided Therapy; CBT4CBT
MeSH Terms: conditions — Alcohol Drinking; Suicidal Ideation; Behavior; Suicide | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alcohol-Based Computer Based Training for Cognitive Behavioral Therapy (Experimental): Participants in this arm will complete four assessments, one at baseline, then another three one month apart. Participants will be given access to Computer Based Training for Cognitive Behavioral Therapy (CBT4CBT) at the end of their baseline session.
  Interventions: Behavioral: Self-Guided Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Self-Guided Cognitive Behavioral Therapy — Computer Based Training for Cognitive Behavioral Therapy (CBT4CBT) is a set of seven modules that consist of different skills trainings that can be accessed by devices with an internet connection. The version of CBT4CBT that will be provided is the alcohol-based CBT4CBT.
  Other Names: Computer Based Training for Cognitive Behavioral Therapy (CBT4CBT)

SUMMARY:
The purpose of this single groups trial is to (Aim 1) determine relationships between alcohol use, suicidal thoughts and behaviors (STBs), and behavioral economic decision-making in a community sample (N = 100) of alcohol using adults who are 18 years of age or older, (Aim 2) is to determine factors that predict engagement with a remote intervention (computer based training for cognitive behavioral therapy; CBT4CBT) for alcohol and its effects on alcohol use, STBs, and decision-making with those same adults.

Participants will complete a baseline assessment and be given access for remote, self-guided CBT4CBT modules for alcohol use. Following this, participants will remotely complete three follow-up assessments over three months. This will allow for determination of incidence and predictors of alcohol use and STBs and determination of predictors of engagement and efficacy of a remote intervention for alcohol use in both samples.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Consume alcohol at least weekly
* A score of 8 or greater on the Alcohol Use Disorder Identification Test (AUDIT)
* Some interest in cutting back on drinking or quitting
* Read and understand English

Exclusion Criteria:

* A score of 31 or greater on the Alcohol Use Disorder Identification Test (AUDIT) at baseline
* Reporting schizophrenia and/or other psychiatric diagnoses other than depression or anxiety at baseline
* Already being in treatment for alcohol use disorder at baseline
* Past month substance use other than cannabis or tobacco

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in Alcohol Use | Assessed at study week 0, 4, 8, and 12
  Participants will complete baseline and remote follow-up assessments. Alcohol use will be measured by timeline follow-back of alcohol use for the previous 4 weeks of time of assessment. General linear mixed-effects modeling will be used to assess changes in alcohol use.
Engagement with Self-Guided Cognitive Behavioral Therapy for Alcohol Use | Assessed at study week 12
  At the end of the study, participant engagement with Computer Based Training for Cognitive Behavioral Therapy (CBT4CBT) modules will be analyzed with ordinary linear regression. Engagement will be defined as the proportion of modules completed.
Change in Suicidal Thoughts and Behaviors | Assessed at study week 0, 4, 8, and 12
  Participants will complete baseline and remote follow-up assessments. Suicidal thoughts and behaviors will be will be measured by the Colombia Suicide Severity Rating Scale. Suicidal ideation severity is measured from a scale of 0 to 25, where higher scores indicate higher levels of suicidal ideation severity. General linear mixed-effects modeling will be used to assess changes in suicidal thoughts and behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Rzeszutek, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data from this study will be made as available as possible either after the end of the funding period or after acceptance for publication, whichever comes first. All shared data will comply with HIPAA guidelines on personally identifiable information.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code